CLINICAL TRIAL: NCT02324335
Title: Phase 2 Study to Evaluate the Efficacy & Safety of Brilacidin Oral Rinse Administered Daily for 7 Weeks in Attenuating Oral Mucositis in Patients With Head & Neck Cancer Receiving Chemoradiation
Brief Title: Study of the Effects of Brilacidin Oral Rinse on Radiation-induced Oral Mucositis in Patients With Head and Neck Cancer
Acronym: Brilacidin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovation Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CTIX-BRI-205
Record Dates: First submitted 2014-12-17; First posted 2014-12-24 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Neoplasms; Mucositis
Keywords: Oral Mucositis; Brilacidin; Chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Stomatitis | interventions — brilacidin; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator Oral Rinse (Placebo Comparator): Water for Injection
  Interventions: Other: Placebo
- Active Comparator Oral Rinse (Active Comparator): Brilacidin 3 mg/mL in Water for Injection
  Interventions: Drug: Brilacidin

INTERVENTIONS:
Drug: Brilacidin — Oral Rinse used 3 times daily for 7 weeks
  Other Names: PMX30063
  Arms: Active Comparator Oral Rinse
Other: Placebo
  Other Names: Water for Injection
  Arms: Placebo Comparator Oral Rinse

SUMMARY:
Oral Mucositis (OM) is a painful and debilitating side effect of many of the drug/radiation regimens used to treat cancer. This study examines the investigational drug brilacidin and its possible application in prevention of oral mucositis in patients undergoing chemoradiation for treatment of head and neck cancer.

DETAILED DESCRIPTION:
This study will examine whether daily oral rinses with a solution containing brilacidin will prevent the occurrences of OM or lessen the severity of OM if it occurs. Patients will use an oral rinse 3 times daily for up to seven weeks during chemoradiation for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to read, understand and sign an informed consent form (ICF)
2. Have recently diagnosed (within previous 6 months) pathologically confirmed, non-metastatic squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or supraglottic larynx that will be treated with CRT therapy as first line non-surgical treatment. Scans (CT, PET, and/or MRI) obtained within 120 days prior to consent for screening can be used to determine the subject's eligibility.
3. Have a plan to receive a continuous course of conventional external beam irradiation delivered by intensity-modulated radiotherapy (IMRT) as single daily fractions of 2.0 Gy to 2.2 Gy with a cumulative radiation dose ≥55 Gy and ≤72 Gy. Planned radiation treatment fields must include at least two oral sites (buccal mucosa, floor of mouth, ventral/lateral tongue, soft palate). [Note: the independent RTQA consultant must confirm that the planned radiation treatment meets the protocol criteria]
4. Have a plan to receive a standard cisplatin chemotherapy regimen administered weekly (30-40 mg/m2) or approximately every 21 days (80-100 mg/m2)
5. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2. However, potential subjects with an ECOG of 3 may be enrolled provided their condition does not preclude performing the actions required by study participation (e.g., opening medication bottles, swishing the oral rinse and spitting out, completing or participating in completion of daily diaries and FACT-H&N forms).
6. Have adequate hematopoietic, hepatic, and renal function at a screening visit
7. Urine or serum pregnancy test: negative for female patients of childbearing potential
8. Agree to utilize medically accepted methods of birth control during study participation and for 90 days following the last treatment with study drug if a female subject is of childbearing potential or if a male subject has an opposite sex partner of child bearing potential.
9. Males or females aged ≥18 years on day of consent.

Exclusion Criteria:

1. Has tumor(s) of the lips, sinuses, salivary glands, nasopharynx, glottic larynx, subglottic larynx or unknown primary tumor
2. Has metastatic disease (M1) Stage IV C
3. Has had prior radiation to the head and neck
4. Plan to be treated with cetuximab (Erbitux®)
5. Planned use of cisplatin as induction chemotherapy.
6. Has a history of other malignant tumors within the last 5 years, except non melanoma skin cancer or in situ cervical carcinoma curatively excised
7. Has had a major surgical procedure, other than for HNC, or significant traumatic injury within 4 weeks prior to the initiation of RT; anticipation of need for major surgical procedure during the course of the study
8. Has incompletely healed sites of dental extractions
9. Has an 12-lead ECG obtained at screening visit which shows medically significant abnormality(ies) (e.g. left bundle branch block, frequent premature ventricular contractions, QTc interval prolongation > 450 msec for males and > 470 msec for females)
10. Has untreated hypertension or has hypertension under treatment that meets protocol definitions.
11. Has active infectious disease undergoing systemic treatment excluding oral candidiasis
12. Has oral mucositis (of any severity) prior to initiation of radiation therapy
13. Has a diagnosis of an immunosuppressive illness or a condition requiring chronic immunosuppression
14. Has known seropositivity for HIV or hepatitis C antibody, or known to be hepatitis B surface antigen positive (testing for these serologic markers is not required for enrollment in this protocol)
15. Use of any investigational agent within 30 days of randomization
16. Is pregnant or breastfeeding
17. Has known allergies or intolerance to brilacidin, cisplatin or carboplatin
18. Has inability to give informed consent or comply with study requirements
19. Has any other condition or prior therapy that in the opinion of the Investigator would make the patient unsuitable for the study and/or unable to comply with requirements for follow-up visits.
20. Is unwilling or unable to agree to swish and spit the study oral rinse three times per day during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Gilbert, Arizona
  - Lakeland, Florida
  - Columbus, Georgia
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Cheektowaga, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Stony Brook, New York
  - Cleveland, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 subjects were randomized, and 59 subjects received study drug; 59 subjects were analyzed for safety, and 46 subjects were analyzed for efficacy.
Groups:
- Placebo Oral Rinse: Water for Injection
  Placebo: Oral Rinse used 3 times daily for 7 weeks
- Active Oral Rinse: Brilacidin 3 mg/mL in Water for Injection
  Brilacidin: Oral Rinse used 3 times daily for 7 weeks
Period: Overall Study
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
Started | 30 | 29
Completed | 21 | 20
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Population: This is the Safety Population. Same as participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Rinse | Active Oral Rinse | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.63) | 60.3 (9.05) | 58.8 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 28 | 21 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severe OM During Radiation Therapy in Subjects Receiving a Cumulative IMRT Dose of at Least 55 Gy
Description: Incidence of severe oral mucositis, defined as grade 3 or 4 on the WHO Oral Mucositis score, experienced during radiation therapy by patients with head and neck cancer receiving a cumulative radiation dose of at least 55 Gy. The higher the score the more severe the mucositis.
Time Frame: 7 weeks
Population: mITT Population included all randomized subjects who received at least one dose of study drug and a cumulative radiation dose of at least 55 Gy (and no more than 72 Gy)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
Number analyzed (Participants) | 25 | 21
Participants
  Severe OM Yes | 15 | 9
  Severe OM NO | 10 | 12

2. Secondary Outcome: Duration of Severe Oral Mucositis (WHO Grade ≥3) [Overall Duration]
Description: Overall duration of severe OM was defined as the number of days from initial WHO Grade ≥3 during radiation therapy to the day prior to the next OM assessment after the last WHO Grade ≥3 during/after radiation therapy.
Time Frame: 11 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
Number analyzed (Participants) | 25 | 21
Days | 3.0 [0 to 52] | 0.0 [0 to 53]

3. Secondary Outcome: Incidence of Severe Oral Mucositis (WHO Grade ≥3) for Subjects Receiving Cisplatin Every 21 Days
Description: Incidence of severe oral mucositis (WHO Grade ≥3) for subjects receiving cisplatin every 21 days
Time Frame: 7 weeks
Population: Subgroup of subjects receiving cisplatin every 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
Number analyzed (Participants) | 14 | 8
Participants
  Severe OM Yes | 10 | 2
  Severe OM NO | 4 | 6

4. Secondary Outcome: Time to Onset of Severe Oral Mucositis (WHO Grade ≥3)
Description: Time to onset of severe oral mucositis (WHO Grade ≥3) analyzed using Kaplan-Meier methods.
Time Frame: 7 weeks
Population: Data is presented for all subjects (censored and uncensored) in the mITT population, with a censored outcome reported as "NA".
Measure: Median (Full Range); unit: days
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
Number analyzed (Participants) | 25 | 21
days | 47 [19 to NA] — Max [censored] 50 days | NA [15 to NA] — Max [censored] 49 days

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time a subject signs the ICF through the End of Study visit (or Early Withdrawal visit for subjects who withdraw or are withdrawn from the study). This could be up to 17 weeks
Description: Non-Serious AEs Treatment Emergent AEs are presented as those events that were experienced by at least 5 (17%) Subjects in any one Treatment Group and with a Difference in Incidence between Groups of at least 3 (10%) Subjects,
Arm/Group | Placebo Oral Rinse | Active Oral Rinse
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 5/30 | 8/29
Other Adverse Events (participants affected / at risk) | 30/30 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Rinse (N=30) | Active Oral Rinse (N=29)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Oral Rinse (N=30) | Active Oral Rinse (N=29)
Fatigue (General disorders) | 13 | 21
Dysgeusia (Nervous system disorders) | 13 | 17
Dry mouth (Gastrointestinal disorders) | 9 | 16
Constipation (Gastrointestinal disorders) | 17 | 13
Oral pain (Gastrointestinal disorders) | 4 | 7
Saliva altered (Gastrointestinal disorders) | 4 | 7
Blood creatinine increased (Investigations) | 3 | 7
White blood cell count decreased (Investigations) | 11 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Headache (Nervous system disorders) | 2 | 6
Blood urea increased (Investigations) | 1 | 6
Radiation skin injury (Injury, poisoning and procedural complications) | 11 | 5
Dizziness (Nervous system disorders) | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 4
Anxiety (Psychiatric disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT02324335/Prot_SAP_000.pdf